CLINICAL TRIAL: NCT04124887
Title: Remineralization Effect of NaF, NaF With TCP, NaF With CPP-ACP, and NaF With CXP Varnishes on Newly Erupted First Permanent Molars: a Randomised Controlled Trial
Brief Title: Remineralization Effect of Fluoride Varnishes on Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Merve Erkmen Almaz, Asist prof, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kırıkkale pedodontics
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Remineralization
MeSH Terms: interventions — Sodium Fluoride; tricalcium phosphate; Phosphates; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sodium fluoride (Active Comparator): Duraphat Varnish containing 5% Sodium fluoride
  Interventions: Drug: Sodium Fluoride
- Tricalcium phosphate (Experimental): Clinpro™ White Varnish containing 5% NaF with TCP
  Interventions: Drug: Tricalcium Phosphate
- Xylitol-coated calcium and phosphate (Experimental): Embrace ™ Varnish containing 5% NaF with CXP
  Interventions: Drug: Xylitol-coated calcium and phosphate
- Casein phosphopeptide amorphous calcium phosphate (Experimental): MI Varnish containing 5% NaF with CPP-ACP
  Interventions: Drug: Casein phosphopeptide amorphous calcium phosphate

INTERVENTIONS:
Drug: Sodium Fluoride — Sodium Fluoride varnish was applied to the targeted teeth at baseline, one and three months.
  Arms: Sodium fluoride
Drug: Tricalcium Phosphate — Varnish with Tricalcium Phosphate was applied to the targeted teeth at baseline, one and three months.
  Arms: Tricalcium phosphate
Drug: Xylitol-coated calcium and phosphate — Varnish with Xylitol-coated calcium and phosphate was applied to the targeted teeth at baseline, one and three months.
  Arms: Xylitol-coated calcium and phosphate
Drug: Casein phosphopeptide amorphous calcium phosphate — Varnish with Casein phosphopeptide amorphous calcium phosphate was applied to the targeted teeth at baseline, one and three months.
  Arms: Casein phosphopeptide amorphous calcium phosphate

SUMMARY:
The aim of this study was to evaluate and compare the efficacy of NaF, NaF with TCP, NaF with CPP-ACP, and NaF with CXP varnishes on newly erupted first permanent molar teeth. The study was carried out in 40 healthy, high caries risk children (DMFS >8), aged six to seven years with newly erupted permanent first molars who referred to the Pediatric Dentistry Clinic of Kırıkkale University Faculty of Dentistry, Kırıkkale, Turkey. A total of 140 teeth were divided randomly into four groups and the varnishes were applied to the determined teeth at baseline, one and three months. The same varnish was used, if there is more than one first molar to be applied of the same patient. The groups were comprised as follows:

Group 1: Duraphat Varnish containing 5% NaF (Colgate-Palmolive, NSW, Australia) (n = 35), Group 2: Clinpro™ White Varnish containing 5% NaF with TCP (3M ESPE, MN, USA) (n = 35), Group 3: Embrace ™ Varnish containing 5% NaF with CXP (Pulpdent, MA, USA) (n = 35), Group 4: MI Varnish containing 5% NaF with CPP-ACP (GC, Tokyo, Japan) (n = 35). All dental treatments of the patients were completed before the varnish application and oral hygiene instructions were given to all children at the start of the study.

Patients were called for follow up appointments at 1, 3 and 6 months, and in the follow-up period DIAGNOdent device (laser fluorescence scanning) was used to monitor mineralization changes. LF measurements were made at baseline (T0), after one month (T1) three months (T2) and six months (T3). Within and between group comparisons were analysed statistically.

ELIGIBILITY:
Inclusion Criteria:

Subject has at least one fully erupted permanent first molar tooth

Exclusion Criteria:

Subject has a permanent first molar tooth with visible cavitation on the tooth surface Subject has a partially erupted permanent first molar tooth.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Monitoring mineralization changes | One, three, six months
  To monitor mineralization changes on permanent first molars, laser fluorescence scanning method was used with DiagnodentPen device.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)